CLINICAL TRIAL: NCT06203184
Title: Effect of Video Game-Based Exercises on Respiratory Muscle Strength and Physical Fitness After Open Heart Surgery
Brief Title: The Effect of Video Game-Based Exercises After Open Heart Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Burcu Bağcı, Director, Sanko University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BurcuB
Record Dates: First submitted 2024-01-02; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Open Heart Surgery; Physical Fitness; Sleep Quality
Keywords: sleep quality; pyhscal fitness; Open Heart Surger; respiratory muscle strenght
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- video game based exercise training (Experimental): Breathing Games; developed by a company called &Breathing Labs&; allow breathing exercises to be implemented based on video games. Studies have reported that breathing exercises accompanied by visual feedback provide additional benefits, and it has been stated that the virtual reality-based approach is an effective method in this respect.
  Interventions: Other: video based exercises
- control group (Other): No intervention will be made to the control group.
  Interventions: Other: video based exercises

INTERVENTIONS:
Other: video based exercises — Respiratory muscle training and other factors will be examined through 12 weeks of video-based game exercises.

SUMMARY:
The aim of the study is to investigate the effects of video game-based exercises applied in addition to the cardiac rehabilitation program applied after open heart surgery, on pulmonary function and functional independence in the acute state.

After ethics committee approval is received; Patients who volunteer to participate in the study will be divided into two groups by simple random method. The first group will be given a 12-week cardiac rehabilitation program after bypass surgery, and the second group will be given video game-based exercise training together with the cardiac rehabilitation program for 12 weeks. It is planned to apply the cardiac rehabilitation program to both groups twice a day during the postoperative period until hospital discharge. The patient's cardiac rehabilitation program after hospital discharge will be carried out in the cardiac rehabilitation unit three days a week. Cardiac r in the video game-based exercise group In addition to rehabilitation; "Breathing Labs Breathing Games" exercises will continue during the hospital stay, and Xbox games will continue after discharge. Evaluations will be made in the preoperative period (within one week before surgery) and at the end of the 12th postoperative week.

DETAILED DESCRIPTION:
Our work; In order to evaluate the effect of video game-based exercises on respiratory muscle strength and physical fitness within the scope of cardiac rehabilitation after open heart surgery; It will be conducted with patients who have undergone open bypass surgery in the Cardiovascular Surgery Department of Private Sani Konukoğlu Training and Research Hospital.

After ethics committee approval is received; Patients who volunteer to participate in the study will be divided into two groups by simple random method. The first group will be given a 12-week cardiac rehabilitation program after bypass surgery, and the second group will be given video game-based exercise training together with the cardiac rehabilitation program for 12 weeks. It is planned to apply the cardiac rehabilitation program to both groups twice a day during the postoperative period until hospital discharge. The patient's cardiac rehabilitation program after hospital discharge will be carried out in the cardiac rehabilitation unit three days a week. Cardiac in the video game-based exercise group In addition to rehabilitation; "Breathing Labs Breathing Games" exercises will continue during the hospital stay, and Xbox games will continue after discharge. Evaluations will be made in the preoperative period (within one week before surgery) and at the end of the 12th postoperative week.

Maximum inspiratory pressure (MIP), maximal expiratory pressure (MEP) with an intraoral pressure measurement device to evaluate the respiratory muscle strength of the patients, Respiratory Function Test to evaluate respiratory function, Sensior Fitness Test to evaluate physical fitness. International Physical Activity Questionnaire - Short Form (IPAQ-SF) to determine the physical activity levels of the cases in daily life, Charlson Comorbidity Index to quantitatively examine the comorbidities that have an impact on prognosis, and to measure the severity of anxiety and depression in cases with physical diseases. Hospital Anxiety and Depression Scale to monitor patients; quality of life and changes, EQ-5D scale to evaluate patients; quality of life, KATZ scale to evaluate independence in daily living activities, Visual Analog Scale to evaluate dyspnea and pain symptoms. , the Pittsburg Sleep Quality Index will be used to evaluate sleep quality, and the Modified Borg Scale will be used to determine exercise intensity.

ELIGIBILITY:
Inclusion Criteria:

* Those who are younger than 65 years old

  * Having undergone open heart surgery
  * Hemodynamically stable
  * At ambulatory level
  * Agreeing to participate in the study
  * Scoring 25 or more from the Mini-Mental Test

Exclusion Criteria:

* • Those diagnosed with previous cerebrovascular accident

  * Those with orthopedic problems that prevent walking
  * Those with uncontrolled diabetes
  * Those with uncontrolled hypertension
  * Those with severe vision problems
  * Having other diseases (pulmonary, neurological, metabolic, etc.) that limit participation in exercise training.
  * Having verbal and/or auditory cooperation problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
tiredness | 12 weeks
  Modified Borg Scale
Comorbid disease status | 12 weeks
  Charlson Comorbidity Index
Hospital Anxiety and Depression | 12 weeks
  Hospital Hospital Anxiety and Depression Scale
Physical Activity | 12 weeks
  International Physical Activity Questionnaire-Short Form (IPAQ-SF)
Measures quality of life status | 12 weeks
  EQ-5D-3l quality of life scale
activity of daily living | 12 weeks
  KATZ İndex
measures pain intensity | 12 weeks
  Visual Analog Scale
Sleep Quality | 12 weeks
  Pittsburg Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: burcu bağcı, Principal Investigator — Sanko University
Locations (1):
- Sanko University, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No